CLINICAL TRIAL: NCT03137290
Title: Comparison Between the Efficacy of Neostigmine Versus Sugammadex Reversal of Rocuronium Induced Neuromuscular Blockade In Paediatric Patients.
Brief Title: Comparing Reversal With Neostigmine and Sugammadex in Paediatric
Acronym: JS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Doctor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JEPeM/281.3(3)
Record Dates: First submitted 2017-04-16; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Neuromuscular Blockade
Keywords: Paediatric general anaesthesia; Rocuronium; Neostigmine; Sugammadex
MeSH Terms: interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neostigmine (Active Comparator): 1 mg of Atropine (1ml) was mixed with 2.5mg of Neostigmine (1ml) and diluted into 10mls with Normal Saline 0.9% in a 10ml standard syringe.
  Interventions: Drug: Neostigmine
- Sugammadex sodium (Experimental): 100mg Sugammadex (1ml) is diluted into 10mls in a standard 10mls syringe with Normal Saline 0.9%.
  Interventions: Drug: Sugammadex Sodium

INTERVENTIONS:
Drug: Neostigmine — The TOF Watch Sx, and Paediatric Bispectral Index (BIS) monitoring were put on patient. Gaseous induction, with oxygen and Sevoflurane was given until BIS was 40-50, then a intravenous line was obtained. 2 mcg/kg of fentanyl was given for analgesia. then,the TOF Watch Sx was calibrated.The patient was paralyzed with 0.6mg/kg of rocuronium, and intubation of the trachea was done once TOF count was less than 1. A maintenance of 0.2 mg/kg of Rocuronium was given boluses every 30 minutes to maintain TOF count between 2-3. At the end of surgery, TOF count was checked to ensure it was between 2-3. Then a reversal dose for TOF count of 2 to 3 was 0.05 mg/kg of Neostigmine with 0.02 mg/kg of Atropine. Therefore the volume would be 0.2 mls per kg is to be administered.
  Other Names: Prostigmine
  Arms: Neostigmine
Drug: Sugammadex Sodium — The TOF Watch Sx, and Paediatric Bispectral Index (BIS) monitoring were put on patient. Gaseous induction, with oxygen and Sevoflurane was given until BIS was 40-50, then a intravenous line was obtained. 2 mcg/kg of fentanyl was given for analgesia. then,the TOF was calibrated.The patient was paralyzed with 0.6mg/kg of rocuronium, and intubation of the trachea was done once TOF count was less than 1. A maintenance of 0.2 mg/kg of Rocuronium was given boluses every 30 minutes to maintain TOF count between 2-3. At the end of surgery, TOF count was checked to ensure it between 2-3. Then the dose for reversal of sugammadex with a TOF count of 2 or 3 would be 2 mg/kg. This will also be equivalent to a volume of 0.2 mls per kg and given at the end of surgery.
  Other Names: Bridion
  Arms: Sugammadex sodium

SUMMARY:
A reversal agent is commonly given to improve neuromuscular function after intra-operative administration of non-depolarizing neuromuscular blocking agents. The administration of conventional reversal agent neostigmine is associated with many undesirable side effects. For almost a decade, a new novel drug sugammadex has been used to specifically antagonize the effect of aminosteroidal neuromuscular blocking agents.

A total of 80 paediatric patients planned for general anaesthesia were divided into two groups and were given either neostigmine+atropine, or sugammadex for reversal once the operation had completed.

DETAILED DESCRIPTION:
RESEARCH HYPOTHESIS

1. Sugammadex has a shorter recovery time (from TOF count of 2 or 3 to TOF ratio of more than 0.9) as compared to neostigmine.
2. Sugammadex has a more stable haemodynamic profile as compared to neostigmine when used to reverse rocuronium induced neuromuscular blockade in paediatric patients.
3. Sugammadex causes less complications or side effects when used in paediatric patients as a reversal for rocuronium induced neuromuscular blockade when compared to neostigmine.

This study was a prospective, double blinded, randomized control study involving 80 selected paediatric patients undergoing various surgeries under general anaesthesia in the operation theatre of Hospital University Sains Malaysia (USM), Kubang Kerian.

Sample size The sample size for this study was calculated using Power and Sample Size Calculation Programme Version 3.0.10.software based on different each respective objectives.

1. To compare the recovery time from Train of four (TOF) count of 2 or 3 to TOF ratio of more than 0.9 between neostigmine and sugammadex in reversal of rocuronium induced neuromuscular blockade in paediatric patients.

   • For objective 1, 33 participants in each respective groups are needed to detect the difference of 8 minutes (480 seconds) in time taken to achieve TOF ratio of 0.9 post-administration of reversal agent (SD was 590, according to Olzem Sacan et al) with 90% power, alpha 0.05. 20% is added for drop out participant. Therefore sample size, n = 33 + (0.2 x 33) = 40 patients.
2. To compare the haemodynamic changes between neostigmine and sugammadex in reversal of rocuronium induced neuromuscular blockade in paediatric patients.

   * For objective 2 (referring to blood pressure), 22 participants in each respective groups are needed to detect the difference of 10 mmHg in mean arterial blood pressure 5 minutes post-administration of reversal agent (SD was 10, according to Olzem Sacan et al) with 90% power, alpha 0.05. 20% is added for drop out participant. Therefore sample size, n = 22 + (0.2 x 22) = 26 patients.
   * For objective 2 (referring to heart rate), 22 participants in each respective groups are needed to detect the difference of 8 beats per minute in heart rate, 5 minutes post-administration of reversal agent (SD was 8, according to Olzem Sacan et al) with 90% power, alpha 0.05. 20% is added for drop out participant. Therefore sample size, n = 22 + (0.2 x 22) = 26 patients.

Therefore the total patients in each group will be 40 patients per group. Total sample size is 80 patients.

After gaining approval from USM Research Ethics Committee, the study was conducted in the Operation Theatre Hospital University Sains Malaysia (HUSM).

Parents of patients who fulfilled the inclusion criteria for this study were counselled, and those who agreed to participate in the study were given full explanation about the study and written consent was taken.

Randomization Subjects were divided into two groups using allocation sequence generated from online randomisation software (http://www.randomization.com). These respective allocations were concealed in sealed envelopes, which were not opened until it was time to administer the respective reversal agents in the Operation Theatre after completion of surgery. Patients were randomised to receive either 'Drug A' or 'Drug B' to reverse rocuronium induced neuromuscular blockade.

The randomization generated by the computer was only known to the anaesthetic assistant nurse, who is not involved in recruiting patients or carrying out the study.

Blinding This is a double blinded study. There were 2 important measures taken to ensure this. For this purpose, a specific anaesthetic assistant nurse is allocated before the study was carried out. This nurse is not involved in recruiting the subjects or carrying out the study, and is not related to the researcher.

Step 1 : Prior to sample collection, all subjects have already been randomized according to a sequence derived from online computer randomization. The anaesthetic assistant nurse prepares 80 envelopes, each respectively numbered 1-80, and 80 cards that will fit into the envelope, 40 labelled 'A' and 40 labelled 'B'. The cards were inserted into the envelopes and sealed according to the sequence that was derived from computer randomization. For example if subject 1 falls under group A, the card labelled 'A' is inserted into the envelope labelled 1, and firmly sealed. This is continued until all 80 cards have been inserted into all 80 numbered envelopes according to the determined sequence, all being firmly sealed. This process is carried out without the presence of the researcher.

Step 2 : On the day of surgery, prior to inducing the patient under general anaesthesia, the anaesthetic assistant nurse had prepares the reversal agents labelled 'Drug A' and 'Drug B'. To ensure desired double blinding, both reversal agents had to be diluted into similar volumes for equivalent dose for each respective drug for reversal of moderate block of Rocuronium induced neuromuscular blockade (TOF count 2 or 3)

* 1 mg of Atropine (1ml) was mixed with 2.5mg of Neostigmine (1ml) and diluted into 10 mls with Normal Saline 0.9% in a 10ml standard syringe. This would be a solution of 0.1 mg/ml Atropine with 0.25 mg/ml Neostigmine. A normal standard reversal dose for TOF count of 2 to 3 would be 0.05 mg/kg of Neostigmine with 0.02 mg/kg of Atropine. Therefore the volume would be 0.2mls per kg.
* 100 mg Sugammadex (1ml) is diluted into 10mls in a standard 10mls syringe with Normal Saline 0.9%. This will provide a new solution of 10mg/ml. The required dose for reversal of reversal of Rocuronium induced neuromuscular blockade with a TOF count of 2 or 3 would be 2mg/kg. This will also be equivalent to a volume of 0.2mls per kg.

This process was also done without the presence of the researcher. All medications were discarded by the end of the day.

Only the anaesthetic assistant nurse is aware which drug, either Neostigmine-Atropine combination or Sugammadex belongs to either group A (drug A) and group B (drug B), till all 80 samples have been collected. After completion of the study, the researcher is informed which drug was labelled as 'Drug A' and 'Drug B' respectively.

Study Protocol In the operating room, the patient was put under routine monitoring for general anaesthesia, including non-invasive blood pressure, electrocardiography, pulse oxymetry, end tidal carbon dioxide. The TOF Watch Sx, was also placed at the patients hand appropriately along the ulnar groove to monitor the neurotransmission activity of ulnar nerve . TOF reading was not taken at this time.

Paediatric Bispectral Index (BIS) monitoring was also placed on the patient's forehead, to ensure the patient was adequately induced prior to any painful stimulation for example intravenous access placement or TOF monitoring.

The patient was induced via sevoflurane gaseous induction, with a fresh gas flow rate of 8 litres per min of oxygen. Sevoflurane was dialled between 4 to 6 percent, to ensure hemodynamic parameters were within acceptable range, and BIS count achieved was 40-50.

Once the patient was fully relaxed and induced, a good functioning appropriate sized peripheral intravenous access was obtained.

2 mcg/kg of fentanyl was given for analgesia. After administration of fentanyl, the TOF Watch Sx was calibrated and a baseline TOF reading was taken and recorded.The patient was paralyzed with 0.6 mg/kg of rocuronium, and intubation of the trachea was done once TOF count was less than 1.

TOF monitoring was assessed at 15 minute intervals once patient was under general anaesthesia. Boluses of intravenous rocuronium 0.2 mg/kg was administered intermittently to maintain a TOF count of 2-3.

The baseline haemodynamic values (blood pressure, heart rate, pulse oxymetry, end tidal carbon dioxide) were documented prior to induction, post-intubation and the subsequent 15 minutes interval, to obtain a baseline and mean reading. The TOF readings were documented prior to Rocuronium administration (post-induction), post-intubation, then every 15 minutes interval, and just prior to reversal.

All patients were given suppositories paracetamol 20-30mg/kg for analgesia. No further opioids were served other than on induction. Where applicable, regional blocks or local infiltration at the surgical site were given for analgesia.

Prior to administration of the reversal agent as determined by randomization, it was ensured that the TOF reading was 2-3.

The following time was taken and recorded :

* from administration of reversal agent to TOF ratio more than 0.9
* from administration of reversal to spontaneous ventilation
* from administration of reversal to adequate ventilation (tidal volume at least 6mls/kg and adequate respiratory rate for age)
* from administration of reversal to extubation The haemodynamic parameters (blood pressure, heart rate, pulse oxymetry, respiratory rate, tidal volume, end tidal carbon dioxide) were documented in 5 minute intervals upon administration of the reversal agent.

Haemodynamic parameters in the recovery bay (blood pressure, heart rate, pulse oxymetry, respiratory rate) were also documented.

Patients were also observed for any complications or side effects post-extubation such as nausea, vomiting, secretions, respiratory distress, etc in the recovery bay.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologist (ASA) physical status 1 and 2.
* Paediatric patients within the above criteria whom require rocuronium induced neuromuscular blockage for general anaesthesia

Exclusion Criteria:

* Active or recent upper respiratory tract infection (within 2 weeks)
* Haemodynamically unstable patients for example trauma, haemorrhage, sepsis, thyrotoxic or cardiac failure
* Patients with pre-existing neuromuscular disorders
* Patients with renal failure, with creatinine clearance of less than 30mmol/L
* Patients requiring post-operative ventilation
* Patients with known allergy to sugammadex or neostigmine

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Recovery time | From the time the reversal drugs (neostigmine or sugammadex) were given at TOF count of 2-3 till the TOF ratio is more than 0.9 up to 5 minutes after the operation finished
  To assess the recovery time from TOF count of 2 or 3 to TOF ratio of more than 0.9 between neostigmine or sugammadex in reversal of rocuronium induced neuromuscular blockade in paediatric patients.

SECONDARY OUTCOMES:
Adequate ventilation | From the time of the reversal drugs (neostigmine or sugammadex) were given till patient achieved good ventilation (tidal volume 6 ml/kg) up to 5 minutes after the operation finished
  To evaluate the time from administration of reversal to adequate ventilation (tidal volume at least 6mls/kg and adequate respiratory rate for age)
Extubation time | From the time of the reversal drugs (neostigmine or sugammadex) were given till the patient is extubated up to 5 minutes after the operation finished.
  To evaluate the time from administration of reversal to extubation
Blood Pressure | From the time of the reversal drugs (neostigmine or sugammadex) were given till the patient is discharged throughout the time the patient stays at the recovery bay up to 30 minutes.
  Blood pressure was documented in 5 minute intervals upon administration of the reversal agent and in the the recovery bay.
Heart Rate | From the time of the reversal drugs (neostigmine or sugammadex) were given till the patient is discharged throughout the time the patient stays at the recovery bay up to 30 minutes.
  Heart rate was documented in 5 minute intervals upon administration of the reversal agent and in the the recovery bay.
Oxygen saturation | From the time of the reversal drugs (neostigmine or sugammadex) were given till the patient is discharged throughout the time the patient stays at the recovery bay up to 30 minutes.
  Oxygen saturation was documented in 5 minute intervals upon administration of the reversal agent and in the the recovery bay.
Number of patients with treatment related-adverse event as assessed by clinical observation | From the time of the patient extubated until the patient is discharged throughout the time the patient stays at the recovery bay up to 30 minutes.
  To monitor any incidence of treatment related-adverse event post extubation

CONTACTS AND LOCATIONS:
Overall Officials: Rhendra Hardy Mohamad Zaini, MD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blobner M, Eriksson LI, Scholz J, Motsch J, Della Rocca G, Prins ME. Reversal of rocuronium-induced neuromuscular blockade with sugammadex compared with neostigmine during sevoflurane anaesthesia: results of a randomised, controlled trial. Eur J Anaesthesiol. 2010 Oct;27(10):874-81. doi: 10.1097/EJA.0b013e32833d56b7. PMID 20683334
- [Result] Khuenl-Brady KS, Wattwil M, Vanacker BF, Lora-Tamayo JI, Rietbergen H, Alvarez-Gomez JA. Sugammadex provides faster reversal of vecuronium-induced neuromuscular blockade compared with neostigmine: a multicenter, randomized, controlled trial. Anesth Analg. 2010 Jan 1;110(1):64-73. doi: 10.1213/ane.0b013e3181ac53c3. Epub 2009 Aug 27. PMID 19713265
- [Result] Plaud B, Meretoja O, Hofmockel R, Raft J, Stoddart PA, van Kuijk JH, Hermens Y, Mirakhur RK. Reversal of rocuronium-induced neuromuscular blockade with sugammadex in pediatric and adult surgical patients. Anesthesiology. 2009 Feb;110(2):284-94. doi: 10.1097/ALN.0b013e318194caaa. PMID 19194156
- [Result] Sacan O, White PF, Tufanogullari B, Klein K. Sugammadex reversal of rocuronium-induced neuromuscular blockade: a comparison with neostigmine-glycopyrrolate and edrophonium-atropine. Anesth Analg. 2007 Mar;104(3):569-74. doi: 10.1213/01.ane.0000248224.42707.48. PMID 17312210